CLINICAL TRIAL: NCT04685187
Title: Validity and Reliability Study of Turkish Adaptation of The Disease Perception Scale in Rheumatic Diseases
Brief Title: Perception of Illness Turkish Validity and Reliability Study
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Collaborators: Akdeniz University (Other); Ondokuz Mayıs University (Other); Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, ASST. PROF., Pamukkale University
Other Study IDs: ONDOKUZMAYISU
Record Dates: First submitted 2020-12-15; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Perception of Disease
Keywords: rheumatic diseases, perception of illness
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In chronic diseases such as rheumatic diseases, it is important to direct the treatment of the disease and to evaluate the disease perception in terms of the course of the disease. As a result of this study, this questionnaire, which will help us gain information about the perception of the disease specific to rheumatic diseases, will be translated into Turkish.

DETAILED DESCRIPTION:
Disease perception is the cognitive aspect of the disease state. Although they experience the same disease in a certain period of their lives, the methods of meeting the disease and coping with the disease differ. Patients try to explain their illnesses in the light of their personal experiences, knowledge, values, beliefs and needs. People create cognitive models to explain and predict events in the outside world. Patients also develop similar patterns of symptoms of transient or long-term disease. Leventhal et al. suggested that patients formed their own coping mechanisms with these cognitive models and developed the self-regulation theory. According to this theory, people create schemas about illness and life-threatening situations in their minds with the information presented to them from concrete and abstract sources. These cognitive models also include beliefs about treatment and control of the condition.

The World Health Organization (WHO) has classified more than 200 musculoskeletal diseases, the most common being rheumatoid arthritis and osteoarthritis. The biopsychosocial model has been drawing attention in rheumatological rehabilitation in recent years. This model acknowledges that the experiences and symptoms of the disease are affected by biological, psychological and social factors. The dysfunction is not only related to the severity of the disease, but also to how the disease is perceived. The patient's beliefs and perceptions about his illness show how the illness affects him both physically and emotionally. Disease perception is based not only on symptoms but also on disease-related consequences, concerns, and past illness experiences of the patient. Recent studies emphasize the importance of disease perception in explaining the difference in treatment outcomes in chronic diseases, including rheumatic diseases.

It was planned to determine the validity and reliability of the Disease Perception Scale in Rheumatic Diseases due to the importance of treatment in rheumatic diseases and the evaluation of disease perception in terms of the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer.
* To be diagnosed with any of the rheumatic diseases (Rheumatoid Arthritis, Spondyloarthropathies, Fibromyalgia, Reactive Arthritis, Sjögren Syndrome, Systemic Lupus Erythematosus) by a specialist.

Exclusion Criteria:

* Being diagnosed with a chronic disease other than rheumatic disease that requires regular medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis, Spondyloarthropathies, Fibromyalgia, Reactive Arthritis, Sjögren Syndrome, Systemic Lupus Erythematosus
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
1) Health Assessment Questionnaire (HAQ) | The first test is made when the patient is directed by the physician. Seventh day after test, re-test is made. For test-retest, the questionnaire will be repeated 7 days apart.
  HAQ has sub-sections that evaluate the inadequacy index (20 questions), pain (one question) and global health status (one question). The last week is questioned in the survey.There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2.
2) Nottingham Health Profile | The first test is made when the patient is directed by the physician. Seventh day after test, re-test is made. For test-retest, the questionnaire will be repeated 7 days apart.
  Nottingham Health Profile (NHP) is a measurement tool that evaluates the health problems of individuals and how these problems affect their daily activities.The questionnaire is divided into two parts. The first parts comprises 38 questions in six categories: sleep, physical mobility, energy, pain, emotional reactions, and social isolation. This first section is weighted to reflect how severe an impact the respondent thinks their health is having on the above areas of life. The second part of the NHP is made up of seven statements about areas of life that are commonly affected by health: paid employment, jobs around the house, social life, personal relationships, sex life, hobbies and interests, and holidays. Scores on the NHP can range from 0 i.e. no distress to 100 i.e severe distress.
Rheumatic Disease Illness Perception Questionnaire | The first test is made when the patient is directed by the physician. Seventh day after test, re-test is made. For test-retest, the questionnaire will be repeated 7 days apart.
  It is a questionnaire consisting of 11 questions that evaluates the cognitive and emotional perception of the disease in individuals with rheumatic disease. The cause and consequences of the disease, the extent to which the patient understands his / her illness, and the emotional changes in the course of the disease and the disease are questioned.

CONTACTS AND LOCATIONS:
Overall Officials: BİLGE BAŞAKCI CALIK, Assoc. Prof., Study Chair — PAMUKKALE UNIVERTSITY; SABAHAT YAPRAK CETİN, Asst. Prof., Study Chair — Akdeniz University; VELİ ÇOBANKARA, Prof.Dr., Study Chair — Pamukkale University; AYŞE AYAN, Assoc.Prof., Study Chair — ANTALYA EDUCATION RESEARCH HOSPITAL
Locations (1):
- Mine Pekesen Kurtca, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We would like to share study protocol and statistical analysis (SAP).

REFERENCES:
- [Background] Llewellyn CD, McGurk M, Weinman J. Illness and treatment beliefs in head and neck cancer: is Leventhal's common sense model a useful framework for determining changes in outcomes over time? J Psychosom Res. 2007 Jul;63(1):17-26. doi: 10.1016/j.jpsychores.2007.01.013. PMID 17586334
- [Background] Petrie KJ, Weinman J. Why illness perceptions matter. Clin Med (Lond). 2006 Nov-Dec;6(6):536-9. doi: 10.7861/clinmedicine.6-6-536. No abstract available. PMID 17228551
- [Background] Lochting I, Fjerstad E, Garratt AM. Illness perceptions in patients receiving rheumatology rehabilitation: association with health and outcomes at 12 months. BMC Musculoskelet Disord. 2013 Jan 16;14:28. doi: 10.1186/1471-2474-14-28. PMID 23324450